CLINICAL TRIAL: NCT03763331
Title: Home-based Leg Heat Therapy for Patients With Symptomatic Peripheral Arterial Disease
Brief Title: Home-based Leg Heat Therapy
Acronym: HHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Roseguini, Bruno, PhD (Individual)
Responsible Party: Principal Investigator, Raghu Motaganahalli, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1801755556
Record Dates: First submitted 2018-11-23; First posted 2018-12-04 (Actual); Results first posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Diathermy

STUDY DESIGN:
Intervention Model Description: Patients were randomized (blocked and stratified by sex) using assignments generated from PROC PLAN in SAS Version 9.4 by the study statistician into one of two groups: those receiving leg heat therapy or those receiving the sham treatment.
Who Masked: Participant
Masking Description: Participants were informed that there were two different categories of heat therapy, "low heat" and "high heat," and that both might be beneficial for claudication symptoms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Sham treatment (Sham Comparator): Participants were dressed in water-circulating trousers that are connected to a pump. Water at 91.4 degrees F was circulated through the pants for 90 minutes daily for 8 weeks..
  Interventions: Device: Control/Sham Treatment
- Heat Therapy (Active Comparator): Participants were dressed in water-circulating trousers that are connected to a pump. Water at 110 degrees F will be circulated through the pants for 90 minutes daily for 8 weeks.
  Interventions: Device: Heat Therapy

INTERVENTIONS:
Device: Control/Sham Treatment — Thermoneutral water will be circulated through water-circulating trousers to maintain skin temperature at baselines levels daily for 90 minutes for 8 weeks.
  Arms: Sham treatment
Device: Heat Therapy — Water at 110 degrees F will be circulated through water-circulating trousers daily for 90 minutes for 8 weeks.
  Arms: Heat Therapy

SUMMARY:
The objective of this study is to evaluate the benefits of participating for 8 weeks in a home-based daily treatment with heat therapy (HT) or a thermoneutral control intervention, as assessed by vascular function, walking tolerance and quality of life.

DETAILED DESCRIPTION:
Heat therapy (HT) is an emerging non-invasive approach that has been shown to enhance vascular function of the leg in old individuals. The objective of this randomized, controlled study is to evaluate the benefits of participating for 8 weeks in a home-based daily treatment with heat therapy (HT) or a thermoneutral control intervention, as assessed by vascular function, walking tolerance and quality of life. The central hypothesis of this study, based on preliminary data, is that exposure to HT will enhance the oxygenation of calf muscles during exercise and as a result, the onset of pain will be delayed and walking performance will be enhanced. The duration (8 weeks) was chosen based on the recent report of Brunt and co-workers that the improvement in endothelial function promoted by repeat HT in sedentary individuals peaks at 8 weeks following the onset of treatment. Heat Therapy will be applied daily for 90 minutes using water-circulating 'pants' connected to a water pump. Outcomes will be assessed at the halfway point (end of week 4), at the completion of the intervention (end of week 8) and 4 weeks after the end of the intervention (week 12).

ELIGIBILITY:
Inclusion Criteria:

* Men and women with a stable symptomatic PAD for ≥6 months
* Ankle brachial index <0.9 in at least one leg
* Age between 40 and 80 years

Exclusion Criteria:

* Uncontrolled Diabetes (HbA1C > 8.5 measured within 3 months prior to date of consent)
* Wheelchair bound
* Use of a walking aid (i.e. cane, crutches, walker, motorized chair)
* Critical limb ischemia (ischemic rest pain or ischemia-related non healing wounds or tissue loss
* Impaired thermal sensation in the legs
* Exercise-limiting comorbidity
* Chronic Heart Failure stages C and stage D (Stage C: structural heart disease is present and symptoms have occurred; Stage D: presence of advanced heart disease with continued heart failure symptoms requiring aggressive medical therapy)
* Morbid obesity BMI > 35 or unable to fit into water-circulating pants
* Open wounds or ulcers on the extremity
* Prior amputation
* Lower extremity revascularization, major orthopedic surgery, cardiovascular event, or coronary revascularization in the previous three months
* Planned revascularization or major surgery during the next six months
* Plans to change medical therapy during the duration of the study
* Active treatment for cancer
* Chronic kidney disease (eGFR <30 by MDRD or Mayo or Cockcroft-Gault formula).
* HIV positive, active HBV or HCV disease.
* Presence of any clinical condition that makes the patient not suitable to participate in the trial.
* Unable to walk on the treadmill

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R Motaganahalli, Principal Investigator — Indiana University
Locations (1):
- IU Heath Methodist, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by referral from the peripheral vascular disease clinic at the Department of Vascular Surgery at Indiana University's Methodist Hospital, the Non-Invasive Vascular Laboratory at Methodist Hospital, and direct participant contact by the Indiana CTSI Research Network (ResNet) office.
  The first participant was randomized on January 14, 2019. Final follow-up occurred on June 21, 2021.
Pre-assignment Details: A total of 542 patients were referred and screened for the study. Four hundred and twenty-eight participants were deemed ineligible and 80 refused to participate. The remaining 34 patients were randomly allocated to receive HT (n = 18) or the control treatment (n = 16).
Groups:
- Sham: Participants will be dressed in water-circulating trousers that are connected to a pump. Water at 33 degrees Celsius will be circulated through the pants for 90 minutes daily for 8 weeks.
- Heat Therapy: Participants will be dressed in water-circulating trousers that are connected to a pump. Water at 43 degrees Celsius will be circulated through the pants for 90 minutes daily for 8 weeks.
Period: Overall Study
Arm/Group | Sham | Heat Therapy
Started | 16 | 18
Completed | 14 | 15
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Non-compliance | 0 | 3

BASELINE CHARACTERISTICS:
Population: Baseline characteristics of participants with PAD that completed the 8-wk intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham | Heat Therapy | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (5.79) | 62.9 (8.9) | 65.9 (7.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 12 | 10 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 12 | 10 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in 6-min Walk Distance
Description: Change in 6-min walk distance from baseline to the 8-week follow-up
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Sham | Heat Therapy
Number analyzed (Participants) | 14 | 15
meters | -0.9 [-5.8 to 14.3] | 21.3 [10.1 to 42.4]

2. Secondary Outcome: Change in Treadmill Peak Walking Time
Description: Change in treadmill peak walking time from baseline to 8-week follow-up
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Sham | Heat Therapy
Number analyzed (Participants) | 14 | 15
seconds | 61.5 (111.2) | 109.5 (85.4)

3. Secondary Outcome: Change in Peak Calf Blood Flow
Description: Change in peak calf blood flow during reactive hyperemia from baseline to the 8-week follow-up
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mL/min/100 g
Arm/Group | Sham | Heat Therapy
Number analyzed (Participants) | 11 | 11
mL/min/100 g | -4.8 (21.9) | -2.8 (11)

4. Secondary Outcome: Change in Leg Cutaneous Vascular Conductance
Description: Change in cutaneous vascular conductance from baseline to the 8-week follow-up
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: percentage of maximal cutaneous vascular
Arm/Group | Sham | Heat Therapy
Number analyzed (Participants) | 14 | 15
percentage of maximal cutaneous vascular | -2.6 (13.9) | -0.7 (16.3)

5. Secondary Outcome: Change in the Vascular Quality of Life Questionnaire-6 Score
Description: Change in Vascular Quality of Life Questionnaire-6 score from baseline to the 8-week follow-up. The total VASCUQOL score is the average score of questions answered and ranges from 1 (worst QOL) to 7 (best QOL)
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham | Heat Therapy
Number analyzed (Participants) | 14 | 15
score on a scale | 0.6 (0.8) | 0.5 (0.6)

6. Secondary Outcome: Change in the Short Form 36 Physical Functioning Score
Description: Change in the physical functioning subscale score from baseline to the 8-week follow-up. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved. A high score defines a more favorable health state.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham | Heat Therapy
Number analyzed (Participants) | 14 | 15
score on a scale | 4.5 (10.8) | 4.5 (15.9)

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study (i.e. approximately 12 weeks).
Arm/Group | Sham | Heat Therapy
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/18
Other Adverse Events (participants affected / at risk) | 0/16 | 4/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham (N=16) | Heat Therapy (N=18)
Supraventricular tachycardia at the onset of treadmill test (Cardiac disorders) | NA | 1 (1) — Supraventricular tachycardia at the onset of treadmill test
Fall during the 6-min walk test (Musculoskeletal and connective tissue disorders) | NA | 1 (1) — Fall during the 6-min walk test
Knee injury (Musculoskeletal and connective tissue disorders) | NA | 1 (1) — Knee injury
Transient mild leg skin irritation (Skin and subcutaneous tissue disorders) | NA | 1 (1) — Transient mild leg skin irritation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-04-10): https://cdn.clinicaltrials.gov/large-docs/31/NCT03763331/Prot_SAP_003.pdf
  • Informed Consent Form (2019-05-23): https://cdn.clinicaltrials.gov/large-docs/31/NCT03763331/ICF_001.pdf